CLINICAL TRIAL: NCT03628638
Title: 2016-11: Blood Sample Collection in Subjects Participating in a Lung Cancer Screening Program
Brief Title: Blood Sample Collection in Subjects Participating in a Lung Cancer Screening Program
Acronym: 2016-11
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-11
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual blood samples may be used for further analysis and future research. Samples may be stored for up to 20 years. These blood samples will be de-identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung Cancer Screening Patients - No Nodules: Subjects in an low dose CT screening program that present no nodules.
  Interventions: Other: Blood Sample Collection
- Lung Cancer Screening Patients - Nodules: Subjects in an low dose CT screening program that present nodules. Additional follow-up data will be collected for up to 12 months and an additional blood sample collected
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Subjects participating in the study will have blood sample collected at enrollment. . For any subjects scheduled for a 12 month follow-up, additional blood samples will be collected at 12 months from enrollment.

SUMMARY:
The primary objective of this study is to establish a control population to assess performance of an investigational diagnostic test targeting lung neoplasms.

DETAILED DESCRIPTION:
Subjects will be participating in a lung cancer screening program at enrollment. Subjects will have a blood sample collected within 60 days of a low-dose CT scan (LDCT). Subjects with nodules present on the LDCT or subjects with a clean LDCT scheduled for a 12-month follow-up may have another blood draw at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, 50 years of age or older.
2. Subject meets one of two lung cancer screening criteria below.

   1. Subject is a candidate for LDCT lung cancer screening and is scheduled for a baseline LDCT scan. There may be circumstances when a patient cannot have an LDCT scan (e.g., due to insurance issues). In these cases, it is allowable for a patient to have a CT scan in order to meet the inclusion criteria. OR
   2. Subject has had previous LDCT scan(s) for lung cancer screening and the most recent LDCT scan prior to enrollment is negative for pulmonary nodules (Lung-RADS category 1, no nodules).
3. Subject understands the study procedures and is able to provide informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Subjects with pulmonary nodules on the most recent LDCT scan prior to enrollment (Lung-RADS category 1 nodules with specific calcifications such as complete, central, popcorn, concentric rings and fat containing nodules are excluded).
2. Prior history of cancer within the past 5 years except for non-melanoma skin cancer.
3. Prior removal of the lung, excluding percutaneous lung biopsy.
4. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be men and women, 50 years of age or older. Subjects will be participating in a lung cancer screening program at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1718 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Biomarker Identification | 27 months
  Biomarkers under evaluation include differential methylation of nucleic acids and altered expression of proteins in blood to detect lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Laura Strong, Study Director — Exact Sciences
Locations (31):
- United States (31):
  - Achieve Clinical Research, Birmingham, Alabama
  - Phoenix Medical Group, Peoria, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - NewportNativeMD, Inc., Newport Beach, California
  - Palmtree Clinical Research, Inc., Palm Springs, California
  - International Research Partners, LLC, Doral, Florida
  - Clinical Trials of Florida, LLC, Miami, Florida
  - Sarkis Clinical Trials, Ocala, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Pasadena Center for Medical Research, Inc., St. Petersburg, Florida
  - UnityPoint Health - St. Luke's Hospital, Cedar Rapids, Iowa
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Lahey Clinic, Inc., Burlington, Massachusetts
  - Boone Hospital Center, Columbia, Missouri
  - Creighton University, Omaha, Nebraska
  - Pulmonary Ultimate Research Experience, LLC, Toms River, New Jersey
  - Northwell Health Physicians Pulmonary Medicine, Manhasset, New York
  - Gotham Cardiovascular Research, PC, New York, New York
  - Clinical Trials Developers, Inc., Milford, Ohio
  - Chest Diseases of Northwestern PA, Erie, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Research Protocol Management Specialists, Pittsburgh, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Anderson Pharmaceutical Research, LLC, Anderson, South Carolina
  - Charleston Research Institution, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Clinical Research of Charleston, Mt. Pleasant, South Carolina
  - South Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Union Pharmaceutical Research, Union, South Carolina
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - ProHealth Care, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after deidentification. This may include text, tables, figures, and appendices. The study protocol, informed consent form, and clinical study report will also be shared.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available from 2 years and ending 4 years after publication. Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research. Data will be available between 2 and 4 years after publication through the Sponsor.